CLINICAL TRIAL: NCT04336202
Title: A Pilot Study of Dose-escalation Strategy of Radiotherapy Followed by Endorectal Brachytherapy With the Use of a New Rectal Applicator in Inoperable, Ederly Rectal Cancer Patients
Brief Title: Watch and Wait Management on Rectal Cancer Patients Using New Swift Local Therapy
Acronym: Whistle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Collaborators: Icad, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Te Vuong, Radiation Oncologist, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2230
Record Dates: First submitted 2020-02-20; First posted 2020-04-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer; Comorbidities and Coexisting Conditions; Inoperable Disease; Brachytherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- External beam radiotherapy + Endorectal brachytherapy (Other): In this study, all participants will receive a treatment of external beam radiotherapy without chemotherapy, which will be followed by three (3) treatments of endorectal brachytherapy with the new applicator.
  Interventions: Radiation: External beam radiotherapy + Endorectal brachytherapy

INTERVENTIONS:
Radiation: External beam radiotherapy + Endorectal brachytherapy — In this study, all participants will receive a treatment of external beam radiotherapy without chemotherapy, which will be followed by three (3) treatments of endorectal brachytherapy with the new applicator.

SUMMARY:
Within our institution, the principal investigator have acquired expertise in endorectal brachytherapy, a localized treatment for colorectal cancer. Until now a modality which uses an endorectal applicator has been used, which has certain limitations. In the context of this study, a new applicator will be used which is already approved by Health Canada for endorectal brachytherapy, thereby improving the participant's quality of life and optimizing treatment time.

DETAILED DESCRIPTION:
The main goal of this study is to treat patients using external beam radiotherapy followed by endorectal brachytherapy using a new applicator. Validating the feasibility of this new applicator, assessing the treatment time required when using it, the necessary workload required and ultimately avoid the need for surgery are our main priorities. Currently, this option is still experimental, although several patients have been treated with this method during the last ten years.

In this pilot study, 45 patients will be recruited, whom have medical conditions (co-morbidities) that make surgery very difficult, or patients that are refusing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis by proctoscopic biopsy of invasive rectal adenocarcinoma will be considered for entry in this study.
* Patient in whom the diagnosis of invasive rectal cancer has been obtained by incisional biopsy (surgical or endoscopic biopsy) that the majority of the tumor has not been removed .
* The tumor should be either palpable by clinical rectal exam or accessible via a rigid proctoscope, and its proximal border should be located no more than 15 cm from the anal verge.
* Rectal cancer clinically stage as T2-T3 N1+ by MRI or endoscopic ultrasound.
* Tumor of 5 cm or less length, non obstructive
* Patient is not suitable for surgery nor chemotherapy due to medical conditions
* Patient must consent to be in the study and consent form must be signed, witnessed and dated prior to registration .
* Patients must be accessible geographically for follow up.
* Adults older than 18 years of age

Exclusion Criteria:

* Patient with malignant rectal tumors other than adenocarcinoma, i.e, sarcoma, lymphoma, carcinoid, squamous cell, cloacogenic, etc.
* Patient who demonstrate prior to randomization, evidence of free perforation, as manifested by free fluid in the abdomen.
* Patient who are curable by standard of care with either surgery or eligible for the Morpheus study.
* Patient who have received any previous therapy (radiation , chemotherapy) for rectal cancer.
* Patient whose tumor is fixed by clinical examination to surrounding structures, precluding the possibility of adequate surgical resection even with pelvic exenteration.
* Patient with a performance status of 3 or 4.
* Patient with tumor involving the anal canal.
* Patient who are pregnant at the time of randomization.
* Patient with psychiatric or addictive disorders that would preclude obtaining informed consent.
* Patient who have multiple primary tumors involving both the colon and rectum that would preclude them from being classified as having only rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the new device | 2 years post treatment
  To measure the percentage (%) of clinical complete responders versus non-complete clinical responders and compare it to the percentage of an already proven device to determine if the new device can be used to treat rectal cancer patients. The cancer response will be assessed by rectoscopy, biopsy and imaging.
Toxicity using the new device | 2 years post treatment
  Use the CTCAE guidelines to measure the percentage (%) of toxicity (G3 and above) of this novel X-Ray device. All grade 3 post-treatment complications will be reported (Proctitis, rectal bleeding, diarrhea). The toxicity will be assessed by the clinician during the follow-up visits.
  An early stopping rule for possible severe toxicity during and post treatment toxicity will be used in this study.
  The following early stopping rules will be applied to test the null hypothesis that the proportion of severe toxicity is less or equal to 25 % at 0.05:
  * 3 severe toxicities (G3-4) out of the first 12 evaluable patients or
  * 5 severe toxicities (G3-4) out of the first 22 evaluable patients or
  * 7 severe toxicities (G3-4) out of the first 36 evaluable patients.
Workload | 2 years post treatment
  To evaluate the workload of this modality in regards to time management (the time required to treat patients (pre-treatment and during treatment) and the number of ressources required. The principal investigator will compare it to an already existent equivalent treatment.

SECONDARY OUTCOMES:
Tumor response | At clinical evaluation, 13 weeks since beginning of treatments
  Number of participants (#) that are complete clinical responders
Local control | 2 years post treatment
  Number (#) of participants with Local control assessed during follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Te Vuong, MD, Principal Investigator — Sir Mortimer B. Davis - Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rutten HJ, den Dulk M, Lemmens VE, van de Velde CJ, Marijnen CA. Controversies of total mesorectal excision for rectal cancer in elderly patients. Lancet Oncol. 2008 May;9(5):494-501. doi: 10.1016/S1470-2045(08)70129-3. PMID 18452860
- [Background] Dekker JW, van den Broek CB, Bastiaannet E, van de Geest LG, Tollenaar RA, Liefers GJ. Importance of the first postoperative year in the prognosis of elderly colorectal cancer patients. Ann Surg Oncol. 2011 Jun;18(6):1533-9. doi: 10.1245/s10434-011-1671-x. Epub 2011 Mar 29. PMID 21445672
- [Background] Garant A, Magnan S, Devic S, Martin AG, Boutros M, Vasilevsky CA, Ferland S, Bujold A, DesGroseilliers S, Sebajang H, Richard C, Vuong T. Image Guided Adaptive Endorectal Brachytherapy in the Nonoperative Management of Patients With Rectal Cancer. Int J Radiat Oncol Biol Phys. 2019 Dec 1;105(5):1005-1011. doi: 10.1016/j.ijrobp.2019.08.042. Epub 2019 Aug 30. PMID 31476417
- [Background] Liang LH, Tomic N, Vuong T, Aldelaijan S, Bekerat H, DeBlois F, Seuntjens J, Devic S. Physics aspects of the Papillon technique-Five decades later. Brachytherapy. 2018 Jan-Feb;17(1):234-243. doi: 10.1016/j.brachy.2017.09.016. PMID 29102741
- [Background] Gerard JP, Chapet O, Ramaioli A, Romestaing P. Long-term control of T2-T3 rectal adenocarcinoma with radiotherapy alone. Int J Radiat Oncol Biol Phys. 2002 Sep 1;54(1):142-9. doi: 10.1016/s0360-3016(02)02879-1. PMID 12182984
- [Background] Sun Myint A, Smith FM, Gollins SW, Wong H, Rao C, Whitmarsh K, Sripadam R, Rooney P, Hershman MJ, Fekete Z, Perkins K, Pritchard DM. Dose escalation using contact X-ray brachytherapy (Papillon) for rectal cancer: does it improve the chance of organ preservation? Br J Radiol. 2017 Dec;90(1080):20170175. doi: 10.1259/bjr.20170175. Epub 2017 Nov 10. PMID 28937269